CLINICAL TRIAL: NCT02419989
Title: Prospective Evaluation of a Standardized Approach to Diagnosis (PREDICT) and Treatment (PATIENCE) of Nontuberculous Mycobacteria Disease in Cystic Fibrosis
Brief Title: PATIENCE Trial: Prospective Algorithm for Treatment of NTM in Cystic Fibrosis
Acronym: PATIENCE
Status: Enrolling by invitation | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Jerry A. Nick, M.D., Professor of Medicine, National Jewish Health
Other Study IDs: NTM-OB-17 (PATIENCE PART B)
Record Dates: First submitted 2014-12-09; First posted 2015-04-17 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
Keywords: Nontuberculous Mycobacteria
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples collected may include serum, sputum, whole blood, breath, urine, and NTM isolates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF patients: Male and female subjects with CF age 6 years and older who meet diagnostic criteria for NTM disease through participation in the PREDICT (Part A) study who are being offered NTM treatment.

SUMMARY:
Isolation of nontuberculous mycobacteria (NTM) from the sputum of individuals with CF is an increasingly common finding, and the lack of an evidenced-based approach to treatment of NTM disease has been identified as one of the greatest unmet needs within the CF community. Current evidence predicts that the prevalence of NTM will remain relatively high in the CF population. Approaches to NTM disease treatment differ widely between centers, and expected outcomes are not known. This study is observational and follows current best practices. The study will help define response to treatment, and collect relevant data associated with treatment of NTM disease to build a framework for future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

1. Previous participation in PREDICT and diagnosis of NTM disease for the same species of NTM
2. Intention to treat for NTM disease for M. avium complex or M. abscessus complex
3. Written informed consent (and assent when applicable) obtained from participant or participant's legal representative
4. Signed informed consent to participate in data submission to the CFF Patient Registry
5. Be willing and able to initiate treatment for NTM and to adhere to study procedures in the context of clinical care, and other protocol requirements

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects with CF age 6 years and older with a confirmed diagnosis of NTM disease who are initiating treatment for NTM.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion who adhere to the protocol based on: number of respiratory cultures obtained per year, withdrawals or major deviations from protocol | 12 months following end of antibiotic treatment

SECONDARY OUTCOMES:
Duration and combinations of NTM treatment regimens received | At end of treatment interval
Proportion requiring antibiotic course change due to intolerance or lack of microbiological conversion (i.e. eradication from sputum) | At end of treatment interval
Proportion who complete ≥ 12 months of treatment since first negative culture | At end of treatment interval
Proportion eradicating NTM defined by ≥ 12 months of negative cultures since end of treatment | 12 months following end of treatment
Variability between sites for NTM eradication success | 12 months following end of treatment
Time to treatment discontinuation due to treatment success | 12 months following end of treatment
Clinical outcomes (FEV1, growth parameters, CFQ-R) | 12 months following end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Nick, MD, Principal Investigator — National Jewish Health; Stacey Martiniano, MD, Principal Investigator — Children's Hospital Colorado
Locations (19):
- United States (19):
  - CFF Pediatric Program, University of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - CFF Adult Program, Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - CFF Pediatric Program University of Michigan, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - CFF Pediatric Program, Columbia University, New York, New York
  - CFF Adult Program, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - CFF Adult Program, The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - CFF Pediatric Program Seattle Children's Hospital, Seattle, Washington
  - CFF Adult Program, University of Washington, Seattle, Washington